CLINICAL TRIAL: NCT04578405
Title: Intracorporeal Anastomosis Accelerates Bowel Function in Comparison to Extracorporeal Anastomosis in Laparoscopic Right Hemicolectomy - a Randomized Control Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Michał Pędziwiatr, Professor, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JagiellonianU-6
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Right Hemicolectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal anastomosis (Active Comparator)
  Interventions: Procedure: Extracorporeal anastomosis
- Intracorporeal anastomosis (Experimental)
  Interventions: Procedure: Intracorporeal anastomosis

INTERVENTIONS:
Procedure: Intracorporeal anastomosis — Anastomosis performed totally laparoscopically
  Arms: Intracorporeal anastomosis
Procedure: Extracorporeal anastomosis — Anastomosis performed through a minilaparotomy
  Arms: Extracorporeal anastomosis

SUMMARY:
Both extracorporeal and intracorporeal anastomosis in laparoscopic right hemicolectomy are renowned and performed worldwide. Many observational studies show conflicting results which method is better. This randomized control trial aimed to assess which technique is superior.

ELIGIBILITY:
Inclusion Criteria:

* malignant or benign neoplasm located in right side of the colon

Exclusion Criteria:

* stage IV disease
* conversion
* inflammatory bowel diseases
* corticosteroid intake
* immunodeficiency
* emergency surgery
* neoadjuvant therapy
* no technical possibility to perform either anastomosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Time to first stool | 5 days

SECONDARY OUTCOMES:
Time to first flatus | 5 days
Complications | 30 day
Length of surgery | 1 day
Length of hospital stay | 30 day

IPD SHARING:
Plan to Share IPD: No